CLINICAL TRIAL: NCT02583347
Title: Sleep Disturbance in Patients With End-Stage Renal Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beaumont Hospital (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Claire Kennedy, Clinical Research Fellow, Beaumont Hospital
Other Study IDs: BH-15/36
Record Dates: First submitted 2015-10-14; First posted 2015-10-22 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Renal Failure Chronic Requiring Hemodialysis; Sleep Disorders
MeSH Terms: conditions — Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Vivia Home Hemodialysis System — The cohort of interest is those patients performing nocturnal home hemodialysis using the Vivia Home Hemodialysis System for 8 hours, 5 nights per week

SUMMARY:
Sleep disorders are common in patients who have chronic kidney disease (CKD). Insomnia is reported in up to 50% of patients treated with hemodialysis compared to 12% of a control population. Restless leg syndrome (RLS) and periodic limb movement disorder (PLM) have been described in 30 to 70% of patients with end stage kidney disease (ESKD). Patients with CKD have also been reported to have a very high prevalence of sleep apnoea disorder. Conventional hemodialysis and peritoneal dialysis do not appear to improve sleep disorders in patients with CKD. There is emerging evidence that nocturnal HD can lead to improvements in sleep quality. Transplantation is thought to improve sleep-related disorders in some but not all patients.

Project Aims

The aims of this project were three-fold:

1. To perform detailed assessment of sleep quality in a cohort of Irish patients with ESRD
2. To assess the feasability and tolerability of unattended home PSG and wrist actigraphy as diagnostic tools in this cohort
3. To assess the impact of a change in RRT modality on sleep quality in Irish patients with ESRD

DETAILED DESCRIPTION:
Patients will not selected based on presence/absence of sleep disturbance. Patients will be prioritized for recruitment if they were active on the transplant waitlist or a change in RRT modality is planned.

Patients will be selected for inclusion if they were >16 years old, competent to independently undertake the informed consent process and are currently on RRT or planned to start RRT in the next three months. The following exclusion criteria will be applied: dementia, active malignancy, major psychiatric disorder, home oxygen therapy, CPAP therapy, and regular benzodiazepine use.

Baseline Evaluation

Baseline evaluation includes the following:

* Demographics and clinical parameters including medications and caffeine intake
* Dialysis prescription and adequacy (weekly standardised Kt/V)
* Laboratory data (haemoglobin, iron, phosphate, PTH)
* Subjective sleep quality as measured by Berlin Questionnaire, Epworth Sleepiness Scale, Pittsburgh Sleep Quality Index and International Restless Leg Syndrome Questionnaire
* Quality of Life as assessed by the 36 Item Short Form Survey (SF-36), Beck Depression Index and Centre for Epidemiologic Studies-Depression Scale
* Cognitive assessment as measured by Trail Making Tests 1 & 2, Category Fluency, Controlled Oral Word Association Test and Hopkins Verbal Learning Test
* Unattended home polysomnography set-up up by investigator who was blinded to the results of the above assessments
* Wrist actigraphy for 3-5 continuous days (Philips Respironics Actiwatch 2 System)

Follow-up Evaluation following RRT Modality Change Follow-up evaluation will be performed in the same way as baseline evaluation at three - six months post switch of RRT modality. As the impact of NHHD is of particular interest, follow-up evaluation will be performed at one and six months post switch to NHHD in those patients who switched to NHHD. The follow-up home PSG was performed on an 'on-dialysis' night and an 'off-dialysis' night to evaluate the impact of the nocturnal procedure itself on sleep.

Data Analysis A sleep technician, blinded to the questionnaire results, compiles the PSG analysis and reports in accordance with the American Academy of Sleep Medicine (AASM) manual for the Scoring of Sleep and Associated Events (40). Actigraphy analysis is reported using Philips Respironics Actiwatch Software.

Statistical methods Statistical analysis will be performed using Stata V14 and Prism V6. All p values <0.05 will be considered statistically significant. Mean data and standard deviation data will be analysed using independent samples t-test and repeated measures analysis of variance (ANOVA). Nominal data will be analysed using chi-squared analysis.

Safety & Tolerability Reports were reviewed with a Respiratory Consultant with specialist interest in Sleep Medicine on a regular basis and abnormal results were discussed in detail. If specific therapy is indicated on the basis of the research tests, the treating nephrologist will be informed and a management plan recommended.

ELIGIBILITY:
Inclusion Criteria:

* >16 years old,
* competent to independently undertake the informed consent process
* currently on RRT or planned to start RRT in the next three months.

Exclusion Criteria:

* Patients consuming Benzodiazepine medication
* Patients requiring nasal CPAP for sleep apnoea
* Patients requiring supplemental oxygen
* Patients with dementia, malignancy, or psychiatric disorder

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Sixty consecutive patients will be enrolled in the study over a period of 24 months. Patients were prioritized for recruitment if they were active on the transplant waitlist or a change in RRT modality was planned.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2015-12; Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
The prevalence of sleep disorders in a cohort of patients with advanced CKD/ESRD | 18 months
  from the total sample population of 60

SECONDARY OUTCOMES:
Change in Subjective Sleep Quality following change of RRT modality | 6 months
  Subjective sleep quality based on validated questionnaire
Change in objective sleep quality following change of RRT modality | 6 months
  Objective sleep quality is measured by means of unattended home polysomnography for one night or wrist actigraphy for 3-5 consecutive nights

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Conlon, MB, MHS, Study Director — Beaumont Hospital
Locations (1):
- Beaumont Hospital, Dublin, Ireland

REFERENCES:
- [Background] Roumelioti ME, Brown LK, Unruh ML. The Relationship Between Volume Overload in End-Stage Renal Disease and Obstructive Sleep Apnea. Semin Dial. 2015 Sep-Oct;28(5):508-13. doi: 10.1111/sdi.12389. Epub 2015 May 5. PMID 25940851
- [Background] Loewen A, Siemens A, Hanly P. Sleep disruption in patients with sleep apnea and end-stage renal disease. J Clin Sleep Med. 2009 Aug 15;5(4):324-9. PMID 19968009
- [Background] Hanly P. Sleep disorders and home dialysis. Adv Chronic Kidney Dis. 2009 May;16(3):179-88. doi: 10.1053/j.ackd.2009.02.004. PMID 19393968
- [Background] Mallamaci F, Leonardis D, Tripepi R, Parlongo G, Catalano C, Tripepi G, Castronovo V, Ferini-Strambi L, Zoccali C. Sleep disordered breathing in renal transplant patients. Am J Transplant. 2009 Jun;9(6):1373-81. doi: 10.1111/j.1600-6143.2009.02653.x. Epub 2009 May 20. PMID 19459802
- [Background] Tang SC, Lam B, Lai AS, Pang CB, Tso WK, Khong PL, Ip MS, Lai KN. Improvement in sleep apnea during nocturnal peritoneal dialysis is associated with reduced airway congestion and better uremic clearance. Clin J Am Soc Nephrol. 2009 Feb;4(2):410-8. doi: 10.2215/CJN.03520708. Epub 2008 Dec 31. PMID 19118118
- [Background] Hanly PJ, Pierratos A. Improvement of sleep apnea in patients with chronic renal failure who undergo nocturnal hemodialysis. N Engl J Med. 2001 Jan 11;344(2):102-7. doi: 10.1056/NEJM200101113440204. PMID 11150360